CLINICAL TRIAL: NCT04720716
Title: A Randomized, Open-label, Controlled, Multicenter Phase III Clinical Study to Compare the Effectiveness and Safety of IBI310 Combined With Sintilimab Versus Sorafenib in the First-line Treatment of Advanced Hepatocellular Carcinoma
Brief Title: A Study to Compare the Effectiveness and Safety of IBI310 Combined With Sintilimab Versus Sorafenib in the First-line Treatment of Advanced HCC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIBI310C301
Record Dates: First submitted 2021-01-13; First posted 2021-01-22 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — sintilimab; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sintilimab combined with IBI310 (Experimental)
  Interventions: Drug: IBI310; Drug: Sintilimab
- Sorafenib (Active Comparator)
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: IBI310 — IBI310 IV d1, Q6W
  Arms: Sintilimab combined with IBI310
Drug: Sintilimab — sintilimab IV d1, Q3W
  Arms: Sintilimab combined with IBI310
Drug: Sorafenib — Sorafenib 400mg po
  Arms: Sorafenib

SUMMARY:
This is a randomized, open-label, controlled, multicenter Phase III study to evaluate the effectiveness and safety of IBI310 combined with sintilimab and sorafenib in patients with locally advanced or metastatic HCC who have not previously received systemic therapy, are unsuitable for radical surgical resection or local treatment, or have had progressive disease after surgical resection or local treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically/cytologically confirmed hepatocellular carcinoma, or liver cirrhosis meeting the clinical diagnostic criteria;
2. ECOG performance status score of 0 or 1 point;
3. No systemic antitumor treatment for hepatocellular carcinoma before the first administration;
4. Barcelona Clinic Liver Cancer stage C, or Stage B not suitable for radical surgery and/or local treatment;
5. At least 1 measurable lesion according to RECIST V1.1);
6. Child-Pugh:≤6
7. Adequate organ and bone marrow function.

Exclusion Criteria:

1. With fibrous lamellar hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, cholangiocarcinoma components in tumor tissues.
2. Have a history of hepatic encephalopathy or have a history of liver transplantation.
3. With clinical symptoms requires drainage of pleural effusion, ascites or pericardial effusion.
4. Central nervous system (CNS) metastasis.
5. Uncontrolled high blood pressure, systolic blood pressure >140mmHg or diastolic blood pressure >90mmHg after optimal medical treatment.
6. Local treatment for liver lesions within 4 weeks.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490 (Estimated)
Dates: Start 2021-02-07 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | up to 24 months after randomization
Objective response rate (ORR) | up to 24 months after randomization
  Objective response rate (ORR) in two arms based on RECIST V1.1 by the IRRC

SECONDARY OUTCOMES:
Progression-free survival (PFS) | up to 24 months after randomization
  Progression-free survival (PFS) in two arms based on RECIST V1.1 by the IRRC and investigator
Duration of response(DOR) | up to 24 months after randomization
  Duration of response(DOR) in two arms based on RECIST V1.1 by the IRRC and investigator
Disease control rate(DCR) | up to 24 months after randomization
  Disease control rate(DCR) in two arms based on RECIST V1.1 by the IRRC and investigator
Time to progression(TTP) | up to 24 months after randomization
  Time to progression(TTP) in two arms based on RECIST V1.1 by the IRRC and investigator
Time to response(TTR) | up to 24 months after randomization
  Time to response(TTR) in two arms based on RECIST V1.1 by the IRRC and investigator
The incidence and severity of Treatment-Emergent Adverse Events | up to 24 months after randomization

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan Universtiy Zhongshan Hospital, Shanghai, Shanghai Municipality, China